CLINICAL TRIAL: NCT02561585
Title: Efficacy of Twice Daily Applications of LEO 124249 Ointment 30mg/g for 12 Weeks to Subjects With Alopecia Areata
Brief Title: LEO 124249 Ointment in the Treatment of Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXP-1222
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2019-02

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 124249 (Experimental): LEO 124249 ointment 30 mg/g twice daily
  Interventions: Drug: LEO 124249
- Vehicle (Placebo Comparator): LEO 124249 ointment vehicle twice daily
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: LEO 124249
  Other Names: LEO 124249 Ointment
  Arms: LEO 124249
Other: Vehicle
  Other Names: LEO 124249 Vehicle
  Arms: Vehicle

SUMMARY:
This clinical trial attempts to investigate the efficacy and safety of LEO 124249 ointment in the treatment of alopecia areata and the molecular disease mechanism and biomarkers.

DETAILED DESCRIPTION:
The objectives of this clinical trial are to compare the efficacy of twice-daily topical LEO 124249 30 mg/g ointment with LEO 124249 ointment vehicle for 12 weeks in the treatment of hair loss in subjects with alopecia areata, to evaluate the safety of this treatment, to evaluate hair regrowth, to determine subject quality of life, and to explore disease mechanism and its biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated informed consent after receiving verbal and written information about the clinical trial.
* Subjects with unequivocal clinical diagnosis of moderate to severe scalp alopecia areata (patch type, totalis, universalis), as determined by the (sub) investigator, affecting a minimum of 30% scalp area at Visit 1 (Screening) and Visit 2 (Day 1, baseline).
* Minimum 6 month duration of hair loss at Visit 1 (Screening). No upper limit time limit.
* Subject must accept to not cut hair in the treated scalp areas during the trial.

Exclusion Criteria:

* Females who are pregnant or are breast feeding.
* Current signs of spontaneous hair regrowth.
* Diffuse type alopecia areata.
* Co-existing moderate to severe androgenic alopecia (Norwood-Hamilton stage IV-VI and Ludwig stage II and III)
* Subjects with changed or expected changes in medication for thyroid disease within 6 month before Visit 1 (screening) or during the trial.
* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), chloroquin derivatives, corticosteroids, or any other systemic therapy that in the opinion of the investigator could affect hair regrowth, within 6 weeks prior to randomization (inhaled or intra-nasal steroids corresponding to up to 1 mg prednisone for asthma or rhinitis may be used).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — The Icahn School of Medicine, Mount Sinai Hospital
Locations (2):
- United States (2):
  - Northwestern University, Evanston, Illinois
  - The Icahn School of Medicine, Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of First Subject First Visit: 02-Feb-2016 Date of Last Subject Last Visit: 06-Dec-2016
Pre-assignment Details: A total of 40 participants were screened, 9 participants were screening failures, and the remaining 31 participants were randomized as follows: 20 participants to LEO 124249 ointment 30 mg/g group and 11 participants to LEO 124249 ointment vehicle group.
Groups:
- LEO 124249 Vehicle: LEO 124249 ointment vehicle twice daily
Period: Overall Study
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Started | 20 | 11
Completed | 17 | 6
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 124249 | LEO 124249 Vehicle | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 11 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (14.0) | 32.1 (8.2) | 34.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Alopecia Areata Tool (SALT) Score
Description: The SALT score indicates the sum area of scalp with hair loss and ranges from 0 - 100 (min-max), with higher scores indicating more hair loss. A negative change in SALT score indicates lesser (improvement) hair loss while positive high scores indicate more (worsening) hair loss.
Time Frame: From baseline (Day 1) to Week 12 (Day 84)
Population: The full analysis set (FAS) was defined as all randomized participants who received at least one application of LEO 124249 (20) ointment or LEO 124249 vehicle (11) and had at least one post-baseline efficacy assessment. Only the participants completing Week 12 have been included in the calculation of the change from baseline in the SALT score.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LEO 124249: LEO 124249 ointment 30 mg/g twice daily application
- LEO 124249 Vehicle: LEO 124249 ointment vehicle twice daily application
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 17 | 6
units on a scale | -3.8 (9.3) | -3.4 (17.0)
Statistical Analysis 1: Comparison: LEO 124249 vs LEO 124249 Vehicle; Test type: Superiority; p = 0.97, t-test, 2 sided — t-test in a baseline adjusted linear model; t-test, 2 sided on a 5% level; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-12.05 to 11.65]

2. Secondary Outcome: Summary of Absolute SALT Score
Description: The SALT (Severity of Alopecia Areata Tool) score indicates the sum area of scalp with hair loss and ranges from 0 - 100 (min-max), with higher scores indicating more hair loss.
  Summary of observed values of the absolute SALT score.
Time Frame: At baseline (Day 1), Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: The full analysis set (FAS) was defined as all randomized participants who received at least one application of LEO 124249 (20) ointment or LEO 124249 vehicle (11) and had at least one post-baseline efficacy assessment. Only the participants who attended the individual visits where included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
units on a scale
  Baseline (Day 1) | 67.2 (25.1) | 74.4 (24.3)
  Week 4 (Day 28): number analyzed (Participants) | 18 | 9
  Week 4 (Day 28) | 63.1 (26.7) | 71.0 (25.9)
  Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Week 8 (Day 56) | 62.7 (27.5) | 68.6 (31.2)
  Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Week 12 (Day 84) | 61.2 (28.9) | 66.4 (38.0)

3. Secondary Outcome: Summary of Change in SALT Score
Description: The SALT (Severity of Alopecia Areata Tool) score indicates the sum area of scalp with hair loss and ranges from 0 - 100 (min-max), with higher scores indicating more hair loss. A negative change in SALT score indicates lesser (improvement) hair loss while positive high scores indicate more (worsening) hair loss.
Time Frame: From baseline (Day 1) to Week 4 (Day 28), Week 8 (Day 56), and Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
units on a scale
  Baseline (Day 1) to Week 4 (Day 28): number analyzed (Participants) | 18 | 9
  Baseline (Day 1) to Week 4 (Day 28) | -2.2 (4.4) | 0.0 (1.3)
  Baseline (Day 1) to Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Baseline (Day 1) to Week 8 (Day 56) | -2.5 (7.3) | -1.5 (9.6)
  Baseline (Day 1) to Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Baseline (Day 1) to Week 12 (Day 84) | -3.8 (9.3) | -3.4 (17.0)

4. Secondary Outcome: Summary of Relative Change in SALT Score
Description: as for outcome 3
Time Frame: From baseline (Day 1) to Week 4 (Day 28), Week 8 (Day 56), and Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
percentage change
  Baseline (Day 1) to Week 4 (Day 28): number analyzed (Participants) | 18 | 9
  Baseline (Day 1) to Week 4 (Day 28) | -4.6 (9.0) | -0.3 (2.3)
  Baseline (Day 1) to Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Baseline (Day 1) to Week 8 (Day 56) | -5.6 (17.8) | -5.3 (16.9)
  Baseline (Day 1) to Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Baseline (Day 1) to Week 12 (Day 84) | -7.7 (22.3) | -9.1 (32.5)

5. Secondary Outcome: Percentage of Patients Who Achieve 50% Improvement in the SALT Score
Description: The event of having at least 50% reduction in SALT score at Week 12 (Day 84) as compared to baseline (Day 1)
Time Frame: At Week 12 (Day 84)
Population: The full analysis set (FAS) was defined as all randomized participants who received at least one application of LEO 124249 (20) ointment or LEO 124249 vehicle (11). Only the participants completing Week 12 have been included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 17 | 6
Participants
  Yes | 2 | 1
  No | 15 | 5

6. Secondary Outcome: Hair Length
Description: Hair length measured in millimeters.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
mm
  Week 4 (Day 28): number analyzed (Participants) | 18 | 9
  Week 4 (Day 28) | 12.7 (17.0) | 5.6 (8.4)
  Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Week 8 (Day 56) | 18.2 (21.7) | 10.3 (16.9)
  Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Week 12 (Day 84) | 25.1 (31.8) | 16.3 (23.5)

7. Secondary Outcome: Hair Growth Rate
Description: Change in hair length measured in millimeters per day.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/day
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
mm/day
  Week 4 (Day 28): number analyzed (Participants) | 10 | 9
  Week 4 (Day 28) | 0.4 (0.7) | 0.1 (0.2)
  Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Week 8 (Day 56) | 0.2 (0.3) | 0.1 (0.5)
  Week 12 (Day 84): number analyzed (Participants) | 17 | 5
  Week 12 (Day 84) | 0.3 (0.8) | 0.1 (0.5)

8. Secondary Outcome: Relative Hair Thickness
Description: Thickness relative to participant's normal scalp hair. Relative assessment not applicable for participants with alopecia areata totalis and universalis.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
Participants
  Week 4 (Day 28): number analyzed (Participants) | 11 | 1
  Week 4 (Day 28): Much thinner | 10 | 1
  Week 4 (Day 28): Slightly thinner | 1 | 0
  Week 4 (Day 28): Same thickness | 0 | 0
  Week 8 (Day 56): number analyzed (Participants) | 8 | 2
  Week 8 (Day 56): Much thinner | 6 | 1
  Week 8 (Day 56): Slightly thinner | 1 | 1
  Week 8 (Day 56): Same thickness | 1 | 0
  Week 12 (Day 84): number analyzed (Participants) | 6 | 2
  Week 12 (Day 84): Much thinner | 4 | 1
  Week 12 (Day 84): Slightly thinner | 1 | 1
  Week 12 (Day 84): Same thickness | 1 | 0

9. Secondary Outcome: Hair Type
Description: Hair type being either vellus hair or terminal hair. Hair type is not applicable for participants with alopecia areata totalis and universalis.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
Participants
  Week 4 (Day 28): number analyzed (Participants) | 13 | 3
  Week 4 (Day 28): Terminal hair | 4 | 1
  Week 4 (Day 28): Velus hair | 9 | 2
  Week 8 (Day 56): number analyzed (Participants) | 13 | 3
  Week 8 (Day 56): Terminal hair | 4 | 2
  Week 8 (Day 56): Velus hair | 9 | 1
  Week 12 (Day 84): number analyzed (Participants) | 12 | 3
  Week 12 (Day 84): Terminal hair | 6 | 1
  Week 12 (Day 84): Velus hair | 6 | 2

10. Secondary Outcome: Hair Color
Description: Absolute color of hair. Hair color is not applicable for alopecia areata totalis and universalis.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
Participants
  Week 4 (Day 28): number analyzed (Participants) | 14 | 3
  Week 4 (Day 28): Black | 4 | 1
  Week 4 (Day 28): Blond | 2 | 1
  Week 4 (Day 28): Brown | 3 | 0
  Week 4 (Day 28): Gray | 0 | 0
  Week 4 (Day 28): Red | 0 | 0
  Week 4 (Day 28): White | 5 | 1
  Week 8 (Day 56): number analyzed (Participants) | 14 | 3
  Week 8 (Day 56): Black | 4 | 1
  Week 8 (Day 56): Blond | 1 | 0
  Week 8 (Day 56): Brown | 4 | 0
  Week 8 (Day 56): Gray | 0 | 1
  Week 8 (Day 56): Red | 0 | 0
  Week 8 (Day 56): White | 5 | 1
  Week 12 (Day 84): number analyzed (Participants) | 12 | 3
  Week 12 (Day 84): Black | 4 | 0
  Week 12 (Day 84): Blond | 1 | 0
  Week 12 (Day 84): Brown | 2 | 0
  Week 12 (Day 84): Gray | 0 | 0
  Week 12 (Day 84): Red | 1 | 0
  Week 12 (Day 84): White | 4 | 3

11. Secondary Outcome: Global Assessment of Overall Hair Regrowth Compared to Baseline
Description: Based on standardized photographs
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
Participants
  Week 4 (Day 28): number analyzed (Participants) | 19 | 9
  Week 4 (Day 28): Much worse | 0 | 0
  Week 4 (Day 28): Moderately worse | 1 | 0
  Week 4 (Day 28): Slightly worse | 1 | 1
  Week 4 (Day 28): Unchanged | 15 | 8
  Week 4 (Day 28): Slightly improved | 2 | 0
  Week 4 (Day 28): Moderately improved | 0 | 0
  Week 4 (Day 28): Much improved | 0 | 0
  Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Week 8 (Day 56): Much worse | 0 | 0
  Week 8 (Day 56): Moderately worse | 0 | 1
  Week 8 (Day 56): Slightly worse | 2 | 0
  Week 8 (Day 56): Unchanged | 14 | 5
  Week 8 (Day 56): Slightly improved | 2 | 0
  Week 8 (Day 56): Moderately improved | 0 | 1
  Week 8 (Day 56): Much improved | 0 | 0
  Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Week 12 (Day 84): Much worse | 0 | 1
  Week 12 (Day 84): Moderately worse | 0 | 0
  Week 12 (Day 84): Slightly worse | 2 | 0
  Week 12 (Day 84): Unchanged | 9 | 4
  Week 12 (Day 84): Slightly improved | 5 | 0
  Week 12 (Day 84): Moderately improved | 1 | 1
  Week 12 (Day 84): Much improved | 0 | 0

12. Secondary Outcome: Participant's Global Assessment of Hair Regrowth
Description: The participant will assess the hair regrowth before the investigator does any assessments of hair regrowth.
Time Frame: At Week 4 (Day 28), Week 8 (Day 56) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
Participants
  Week 4 (Day 28): number analyzed (Participants) | 18 | 9
  Week 4 (Day 28): No regrowth | 8 | 6
  Week 4 (Day 28): <25% of regrowth | 8 | 3
  Week 4 (Day 28): 25%-49% of regrowth | 2 | 0
  Week 4 (Day 28): 50%-74% of regrowth | 0 | 0
  Week 4 (Day 28): 75%-99% of regrowth | 0 | 0
  Week 4 (Day 28): 100% of regrowth | 0 | 0
  Week 8 (Day 56): number analyzed (Participants) | 18 | 7
  Week 8 (Day 56): No regrowth | 8 | 5
  Week 8 (Day 56): <25% of regrowth | 8 | 1
  Week 8 (Day 56): 25%-49% of regrowth | 0 | 1
  Week 8 (Day 56): 50%-74% of regrowth | 2 | 0
  Week 8 (Day 56): 75%-99% of regrowth | 0 | 0
  Week 8 (Day 56): 100% of regrowth | 0 | 0
  Week 12 (Day 84): number analyzed (Participants) | 17 | 6
  Week 12 (Day 84): No regrowth | 6 | 3
  Week 12 (Day 84): <25% of regrowth | 8 | 1
  Week 12 (Day 84): 25%-49% of regrowth | 1 | 1
  Week 12 (Day 84): 50%-74% of regrowth | 2 | 1
  Week 12 (Day 84): 75%-99% of regrowth | 0 | 0
  Week 12 (Day 84): 100% of regrowth | 0 | 0

13. Secondary Outcome: Subcategory and Total Score of the Alopecia Areata Quality of Life Questionnaire (AA-QLI)
Description: The scale includes 21 questions measuring the degree to which the patient was affected by the AA in the last month, scored from 1 (not affected at all) to 4 (highly affected).
  The AA-QLI transformed scores for each of the subcategories 'subjective symptoms', 'relationship' and 'objective signs' ranging from (min-max) 9-36, 9-36, and 3-12. Total score ranges from 0-84.
  Low score indicating that the participant was least affected by AA.
Time Frame: At baseline (Day 1) and at Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: LEO 124249; Week 12: LEO 124249: LEO 124249 ointment 30 mg/g twice daily application
- Baseline: LEO 124249 Vehicle; Week 12: LEO 124249 Vehicle: LEO 124249 ointment vehicle twice daily application
Arm/Group | Baseline: LEO 124249 | Baseline: LEO 124249 Vehicle | Week 12: LEO 124249 | Week 12: LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11 | 20 | 11
units on a scale
  Subjective symptoms | 25.9 (4.9) | 24.3 (5.5) | 25.5 (4.4) | 23.7 (7.3)
  Relationship | 18.7 (6.8) | 17.5 (6.7) | 18.7 (7.2) | 16.8 (7.5)
  Objective signs | 7.8 (2.4) | 8.4 (2.2) | 6.9 (2.3) | 7.7 (2.7)
  Total score | 52.3 (12.1) | 50.2 (11.1) | 51.1 (12.5) | 48.2 (15.2)

14. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Score
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM II) is a validated, general measure of treatment satisfaction for medication - accounting for effectiveness, side effects, convenience, and global satisfaction - that is comparable across medication types and patient conditions.
  The individual derived score for each of the 4 dimensions (effectiveness, side effects, convenience, and global satisfaction) of the TSQM II questionnaire ranged from 0-100, with a higher score indicating greater satisfaction to treatment.
Time Frame: At Week 12 (Day 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 124249 | LEO 124249 Vehicle
Number analyzed (Participants) | 20 | 11
units on a scale
  Effectiveness: number analyzed (Participants) | 17 | 6
  Effectiveness | 28.9 (23.2) | 41.7 (12.9)
  Side effects: number analyzed (Participants) | 16 | 6
  Side effects | 94.5 (15.1) | 100.0 (0.0)
  Convenience: number analyzed (Participants) | 17 | 6
  Convenience | 52.3 (17.7) | 54.6 (21.8)
  Global satisfaction: number analyzed (Participants) | 17 | 6
  Global satisfaction | 40.7 (22.6) | 47.2 (22.8)

ADVERSE EVENTS:
Time Frame: From screening (within 28 days prior to Day 1) to end of trial (Week 14)
Description: Treatment emergent adverse events are reported from baseline (Day 1) to end of trial (Week 14). No adverse events was reported prior to Day 1.
Arm/Group | LEO 124249 | LEO 124249 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 5/20 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 124249 (N=20) | LEO 124249 Vehicle (N=11)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No